CLINICAL TRIAL: NCT06427460
Title: Central-boost Ablative Radiation Therapy for Large Tumors or Tumors Adjacent to Organs at Risk
Brief Title: Central-boost Ablative Radiation Therapy for Solid Tumors (CBART)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhang Huo Jun, Professor, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Changhai Hospital NMU
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; stereotactic body radiation therapy; inner gross tumor volume; central boost; ablative radiation dose
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- stereotactic body radiation therapy (Experimental): Central-boost ablative doses delivered by SBRT.
  Interventions: Radiation: Central-boost ablative dose delivered by stereotactic body radiation therapy

INTERVENTIONS:
Radiation: Central-boost ablative dose delivered by stereotactic body radiation therapy — An inner and complete gross tumor volume (iGTV) is created within the gross tumor volume (GTV). For the liver or lung tumor, the convetional radiation dose is 35-45Gy/5f. Regarding the pancreatic tumor or retroperitoneal tumor, the radiation dose is 30-40Gy/5f. Hence, the radiation dose of iGTV should not be less than 120% of the dose of GTV.

SUMMARY:
In the case of large tumors or tumors closely adjacent to organs at risk, ablative doses offered by stereotactic body radiation therapy (SBRT) could not be delivered. Therefore, a technique that could provide high radiation doses to tumors without increasing of risks of severe adverse effects is required.

DETAILED DESCRIPTION:
Regarding the advanced stage tumor, especially tumors with large volumes or closely adjacent to organs at risk, patients are not candidates for surgical resection. Therefore, raduitherapy may be the optimal local therapy to ameliorate symptoms and be combined with systemic therapy, including chemotherapy, targeted therapy or immunotherapy. However, for those tumors, ablative doses could not be given due to large volumes and abutting to organs at risk.

In order to solve the problem, spatially fractionated radiation therapy (SFRT) is used. In details, it was performed based on grid or lattice, which creates several cylindrical high-radiation-dose areas in tumors. Nevertheless, the ablative dose areas are limited albeit with SFRT, which may not greatly improve tumor local. Hence, we create an inner and complete inner gross tumor volume that would be delivered ablative radiation doses, which is named as central-boost ablative radiation therapy (CBART). We aim to investigate the efficacy and safety of CBART in large tumors or tumors adjacent to organs at risk.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years.
* Pathologically confirmed lung, liver, pancreas or retroperitoneal malignant tumor.
* Oligometastasis in the case of metastatic tumor
* the shortest diameter ≥2cm or the distance from the tumor to the organs at risk less than 5mm
* ECOG of 0 to 1 point
* No abnormality in blood routine test, liver and kidney function test and coagulation test (White blood cell count ≥4.0×10^9/L, neutrophil count ≥2.0×10^9, hemoglobin level ≥100g/L, platelet count ≥100×10^9/L, ALT and AST level < 2.5 times the upper limit of normal, total bilirubin and creatinine level within the normal, international normalized ratio <2)

Exclusion Criteria:

* History of radiotherapy for the lesion
* History of tumor within 5 years
* ECOG ≥2 points
* Significant abnormality in blood routine test, liver and kidney function test and coagulation test
* Active inflammatory bowel disease in the case of pancreas or retroperitoneal tumor
* Gastrointestinal bleeding or perforation within 6 months in the case of pancreas or retroperitoneal tumor
* Infections required antibiotics
* Heart or respiratory insufficiency
* Pregnant or breastfeeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2024-05-12 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
One-year local control will be determined. | 1 year
  The proportion of patients without tumor local progression at one year. The progression is assessed by the Response Evaluation Criteria in Solid Tumors (RECIST; version 1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.

SECONDARY OUTCOMES:
Overall survival will be determined. | 2 years
  The time from the enrollment to death.
Progression free survival will be determined. | 2 years
  The time from the enrollment to documentation of any clinical or radiological disease progression or death, whichever occurred first. Progression is assessed by the Response Evaluation Criteria in Solid Tumors (RECIST; version 1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Treatment related adverse events | 2 years
  Treatment-related adverse effects are determined by National Cancer Institute Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Huojun Zhang, M.D., Principal Investigator — Changhai Hospital
Locations (1):
- Huojun Zhang, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No